CLINICAL TRIAL: NCT00498901
Title: Phase II Pilot of Aromatase Inhibitor Therapy With Femara® (Letrozole) and Ovarian Suppression in Premenopausal Estrogen Receptor Positive Women With Stage IV Carcinoma of the Breast
Brief Title: Letrozole and Goserelin or Leuprolide in Treating Premenopausal Estrogen Receptor-Positive Patients With Stage IV Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Hannah M. Linden, University Cancer Center at University of Washington Medical Center
Masking: None | Purpose: Treatment
Other Study IDs: 6412; FHCRC-6412; UWCC-UW 6412; UWCC- 06-4560-H/D; CDR0000553612 (Registry Identifier: pdq)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2013-05-09 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Letrozole; Leuprolide

INTERVENTIONS:
Drug: goserelin
Drug: letrozole
Drug: leuprolide acetate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Aromatase inhibitors, such as letrozole, prevent the formation of estradiol, a female hormone. Giving letrozole together with goserelin, leuprolide, or surgery may be an effective treatment in women with hormone-dependent breast cancer.

PURPOSE: This phase II trial is studying how well giving letrozole together with goserelin or leuprolide works in treating premenopausal estrogen receptor-positive patients with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To measure overall response rate (ORR) in premenopausal women treated with an aromatase inhibitor (AI) and ovarian suppression (OS).

Secondary

* To measure time to treatment failure (TTF) in premenopausal women treated with an AI and OS.
* To measure time to progression (TTP) in premenopausal women treated with an AI and OS.
* To measure time to death in premenopausal women treated with an AI and OS.
* To assess the clinical benefit rate (CBR) in premenopausal women treated with an AI and OS.
* To measure the qualitative and quantitative toxicity of an AI and OS.
* To determine whether ORR, TTP, and CBR are similar to what is seen in postmenopausal women treated with an AI.
* To determine whether ORR, TTP, and CBR are similar to what is seen in premenopausal women treated with tamoxifen and OS.
* To determine if levels of estrogen (i.e., estradiol or estrone) are adequately suppressed in premenopausal women on an AI and OS.

OUTLINE: This is a pilot, open-label study.

Patients undergo surgical ovarian suppression (OS) or medical OS with luteinizing hormone-releasing hormone (LHRH) agonist (i.e., goserelin or leuprolide acetate, intramuscularly once monthly for 3 months and then every 2 months thereafter for the duration of study therapy). Beginning on day 14 after initiation of LHRH-agonist therapy or surgery, patients receive oral letrozole once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Menopausal status is tested periodically during study by measuring serum estradiol levels. Patients not converting to a menopausal state after the first month of study therapy, receive a higher dose of LHRH and undergo repeat estradiol testing in the second month. If the patient continues to be premenopausal, they are then considered for bilateral salpingo-oophorectomy or removed from study.

After completion of study therapy, patients are followed every 3 months for 2 years, every 6 months for 2 years, and annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the breast

  * Metastatic disease
* Measurable disease (i.e., unidimensional by RECIST)
* No rapidly progressing visceral involvement (e.g., liver or lymphangitic lung disease)
* No known marrow involvement as evidenced by diffuse uptake by imaging studies or bone marrow biopsy or aspirate
* No evidence of CNS metastases
* Estrogen- and/or progesterone-receptor positive status confirmed in primary breast tumor or in recent biopsy of metastatic site

PATIENT CHARACTERISTICS:

* Female
* Premenopausal*, as defined by the following criteria:

  * Less than 12 months from last menstrual period or premenopausal estradiol within the past 12 months
  * No prior bilateral oophorectomy
  * 45 years old or younger with intact ovaries and not a candidate for aromatase inhibitor therapy alone due to the potential for recurrent ovarian function NOTE: *Women are considered premenopausal after prior hysterectomy if they have intact ovaries and follicular hormone levels consistent with the institutional normal values for the premenopausal state
* Women meeting premenopausal criteria prior to receiving ovarian suppression are eligible
* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for 12 weeks after discontinuation of study therapy
* ANC ≥ 500 cells/mm³
* Platelet count ≥ 50,000 cells/mm³
* Hematocrit ≥ 28%
* In the absence of liver metastases:

  * AST and ALT ≤ 2.5 times upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2.5 times ULN
* In the presence of liver metastases:

  * AST and ALT ≤ 5 times ULN
  * Alkaline phosphatase ≤ 5 times ULN
* In the presence of bone metastases:

  * AST and ALT ≤ 10 times ULN
  * Alkaline phosphatase ≤ 10 times ULN
* Total bilirubin ≤ 2 times ULN
* No significant comorbid conditions, including any of the following:

  * Clinically significant cardiac disease not well controlled with medication (e.g., congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias)
  * Myocardial infarction within the past 12 months
  * Serious concurrent infection
* No lack of physical integrity of the upper gastrointestinal tract
* No inability to swallow or malabsorption syndrome
* No other carcinoma within the past 5 years except nonmelanoma skin cancer and treated in situ cervical cancer
* No mental illness
* No known hypersensitivity to luteinizing hormone-releasing hormone (LHRH), LHRH-agonist analogues, or any of the components in goserelin

PRIOR CONCURRENT THERAPY:

* No concurrent chemotherapy and/or additional hormonal therapy
* Concurrent trastuzumab (Herceptin®) for patients with HER2 overexpression allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-02; Primary Completion 2007-12 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate as measured by RECIST

SECONDARY OUTCOMES:
Time to treatment failure
Time to progression
Time to death
Clinical benefit rate
Qualitative and quantitative toxicity as assessed by NCI CTCAE v3.0
Disease-free survival
Overall survival
Safety
Comparison of response with results of previous studies of postmenopausal women treated with aromatase inhibitor (AI) therapy and of premenopausal women treated with ovarian suppression (OS) and tamoxifen
Determination of adequacy of estrogen suppression by AI therapy and OS

CONTACTS AND LOCATIONS:
Overall Officials: Hannah M. Linden, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington